CLINICAL TRIAL: NCT02910830
Title: Osteoarthritis Relationships and Tobacco " Ancillary Study Khoala "
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 13-PP-04
Record Dates: First submitted 2016-09-13; First posted 2016-09-22 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Osteoarthrosis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The role of tobacco in osteoarthritis remains controversial. The Khoala cohort is the first multicenter French cohort of subjects with knee and / or hip osteoarthritis prevalent . It guarantees its methodology great representativeness and therefore an interesting material for the study of risk factors in the population. In addition, it should have little here Radiographs of hands for all its patients. It therefore has the opportunity to study a possible relationship between tobacco and hip osteoarthritis , knee and hand but also to study the relationship between tobacco and structural evolution of hip osteoarthritis and / or symptomatic knee.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged between 40 and 75 years
* hip osteoarthritis and / or knee ( stifle ) , unilateral or bilateral , symptomatic with a confirmed diagnosis and meeting the ACR criteria , representative of prevalent cases in France during the constitution of the cohort
* Affiliation to social security

Exclusion Criteria:

* Presence of a hip or knee prosthesis of the painful joint at baseline ;
* Antecedent osteotomy ;
* severe comorbidity likely to affect significantly the quality of life or induce a major healthcare consumption regardless of osteoarthritis ;
* Knee pain with patellofemoral osteoarthritis isolated , that is to say without tibiofemoral osteoarthritis associated ;
* Other pathologies of these joints
* adults subject to a legal protection measure or unable to express their opposition not to participate in the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with osteoarthritis of the hip and patients with knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 848 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
relationship between smoking and severity of functional impairment in patients with osteoarthritis of hip and knee osteoarthritis using datas from cohort KOHALA | 5 years

IPD SHARING:
Plan to Share IPD: No